CLINICAL TRIAL: NCT03633773
Title: Safety and Efficacy Evaluation of MUC-1 CART in the Treatment of Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-Y2018-078
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: ICC; Mucin-1; CAR-T; Immunotherapy
MeSH Terms: conditions — Cholangiocarcinoma; Medullary cystic kidney disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MUC-1 CART (Experimental): Patients are given fludarabine and cyclophosphamide as pretreatment before MUC-1 CART immunotherapy. After treatment, specific antibodies, CART cells and serum levels of cytokines will be assessed.
  Interventions: Biological: MUC-1 CART cell immunotherapy

INTERVENTIONS:
Biological: MUC-1 CART cell immunotherapy — After fludarabine and cyclophosphamide pre-chemotherapy，MUC-1 CART immunotherapy is given. A decent interval later, levels of specific antibodies, CART cells and serum cytokines will be assessed.

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) is one of the most common liver malignancies. Surgical treatment is the first choice. However, for patients without surgical indications, the benefits of conventional chemoradiotherapy are limited. CART is one of the fastest developed treatments in recent years. MUC-1 CART can target abnormal glycosylation of MUC-1 and then killing tumor specifically. Here, investigators intend to evaluate the safety and efficacy of MUC-1 CART in intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Investigators chose MUC-1 positive intrahepatic cholangiocarcinoma patients with one measurable lesion at least. After general assessment, MUC-1 CART treatment was given to the participants. Objective remission rate, disease control rate, duration of overall response, progression-free survival, overall survival, drugs related side effects and other endpoints events were recorded and analyzed, to assess the MUC-1 CART could or couldn't effectively control the progress of intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old.
2. The expression of ST glycosylated MUC-1 was more than 1+ in immunohistochemistry(IHC) by applicant-approved laboratory.
3. Histopathology or cytology confirmed intrahepatic cholangiocarcinoma.
4. Patients who are unable to perform surgery or are not suitable for surgery, or who have recurrence after surgery, or who are unwilling to undergo chemotherapy.
5. With at least one extracranial measurable lesion according to RECIST 1.1 edition.
6. The expected survival time is more than 60 days.
7. The main organs are functional and meet the following criteria:

1) ECOG physical fitness score was 0~1 or KPS score >70. 2) Routine blood tests were in accordance with the following criteria: HB (>90 g/L) (no blood transfusion within 14 days), ANC (>1.5 x10^9/L), PLT (> 80 x10^9/L), lymphocyte (> 0.7 x10^9/L), LY (> 15%), Alb (> 2.8 g/dL), serum lipase and amylase < 1.5^ULN (upper limit of normal value).

3) Biochemical examination should meet the following criteria: TBIL < 1.5x ULN (upper limit of normal value); ALT < 2.5 xULN; serum Cr<1 xULN; endogenous creatinine clearance > 50ml/min (Cockcroft-Gault formula).

4) Cardiac ejection fraction >55%. 8. No active hemorrhagic disease or severe coagulation dysfunction. 9. No allergy to the contrast media. 10. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the results are negative, and are willing to use appropriate contraception methods during the experiment and 8 weeks after the last CART.

11. The volunteers voluntarily joined the study, signed informed consent, and had good compliance and follow-up.

Exclusion Criteria:

1. The transduction efficiency of T cells was <10% or T cells expanded less than 5 times after culture.
2. Chimeric antigen receptor therapy or other transgenic T cell therapy.
3. Pregnant or lactating women.
4. In the first 4 weeks before the start of the study, they took part in other drug clinical trials.
5. Patients with hypertension who can not be well controlled by a single antihypertensive drug (SBP> 140 mmHg, DBP> 90 mmHg), myocarditis or congenital heart disease, myocardial ischemia or infarction above grade I, arrhythmia above grade I (including QT interval < 440 ms) or cardiac insufficiency.
6. Long term unhealed wounds or fractures.
7. With a history of psychotropic substance abuse and unable to quit or have a history of mental disorders.
8. Past and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc.
9. With uncontrollable fungi, bacteria, viruses or other infections, or need antibacterial treatment. The presence of simple urinary tract infections and uncomplicated bacterial pharyngitis is allowed after consultation with a medical supervisor, if there is a response to active therapy.
10. According to the NCI-CTCAE 4.0 standard, the patients who had used chemotherapy in the past had grade 2 hematological toxicity or grade 3 non-hematological toxicity.
11. With a history of HIV or hepatitis B or hepatitis C virus infection.
12. There are any indwelling catheters or drainage tubes (e.g. percutaneous nephrostomy, Frey's catheter, bile drainage or pleural/peritoneal/pericardial catheter). The use of dedicated central venous catheters is permitted.
13. With brain metastases.
14. With a history or disease of CNS, such as epileptic seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving CNS.
15. With a major immunodeficiency.
16. The main therapeutic drugs in this study (including fludarabine, cyclophosphamide, sodium mesylate, tropizumab and anti-infective drugs used during pretreatment) had a history of severe hypersensitivity.
17. In the first 6 months of admission, there was a history of deep venous thrombosis or pulmonary embolism.
18. History of autoimmune diseases (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) that cause terminal organ injury or require systemic immunosuppressive/systemic disease-regulating drugs.
19. With any diseases that may interfere with the safety or efficacy of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | Up to approximately 12 months
  Percentage of patients whose cancer doesn't progress after treatment

SECONDARY OUTCOMES:
Objective response rate | Up to approximately 12 months
  Percentage of patients whose cancer shrinks or disappears after treatment
Duration of overall response | Up to approximately 12 months
  The time of initial response until documented tumor progression.
Progression-free survival | Up to approximately 12 months
  The percentage of people does not get worse for a period of time after diagnosis
Overall survival | Up to approximately 12 months
  The percentage of people still alive for a given period of time after diagnosis
Common Toxicity Criteria for Adverse Effects | Up to approximately 12 months
  According to Common Toxicity Criteria for Adverse Effects version 4
EORTC QLQ - PAN26 | Up to approximately 12 months
  Assessed by the European Organization for Research and Treatment of Cancer Quality of Life
Anti-MUC1 CART cell antibody | Up to approximately 12 months
  Serum level of anti-MUC1 CART cell antibody
MUC1 CART cell | Up to approximately 12 months
  Serum level of MUC-1 CART cell
Related cytokine | Up to approximately 12 months
  Serum level of related cytokine(like IL-2、IL-6、TNF-α、IFNγ and so on)

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided